CLINICAL TRIAL: NCT02048085
Title: A Randomized, Open Label, Pilot Study to Assess the Pharmacodynamics Using Vefiynow and VASP Assay; and Pharmacokinetics of Ticagrelor vs Clopidogrel in Patients Undergoing PCI With History of Fibrinolysis in 24-48 Hours
Brief Title: Comparing Ticagrelor and Clopidogrel Pharmacodynamics After Thrombolysis
Acronym: TACAT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to get study up and enrolling
Sponsor: Medical Center of South Arkansas (Other)
Responsible Party: Principal Investigator, Rakesh K. Sharma, Chief of Medicine, Adjunct Clinical Professor of Medicine and Cardiology, Medical Center of South Arkansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ISSBRIL0224
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction; Acute Coronary Syndrome
Keywords: ACS; STEMI; Fibrinolysis; Pharmacodynamics; Pharmacokinetics; Plavix; Brilinta; Ticagrelor; Clopidogrel
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Acute Coronary Syndrome | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor Arm will be dosed with a loading dose of 180 mg followed by maintenance dose of 90 mg BID until discharge or up to 8 days.
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel arm will be dose with a loading dose of 300 mg followed by maintenance dose of 75 mg everyday until discharge or up to 8 days.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — For ticagrelor arm, randomized STEMI patients with a history of fibrinolysis within last 24-48 and undergoing PCI will be loaded with ticagrelor 180 mg prior to PCI followed by maintenance dose of 90 mg bid.
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Clopidogrel — For clopdigrel arm, randomized STEMI patients with a history of fibrinolysis within last 24-48 and undergoing PCI will be loaded with clopidogrel 300 mg prior to PCI followed by maintenance dose of 75 mg QD
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
This study involves doing platelet function testing in patients who have undergone fibrinolysis. Fibrinolysis (Use of clot busting medicine in heart attack) is the standard of care to restore blood flow in blocked arteries as soon as possible after the "Heart attack" in rural health center where access to cardiac catheterization is one hour away. Fibrinolysis is done by the emergency room physician in a timely fashion to minimize the damage of the myocardium. Additionally anti-platelet regimen as adjuvant for patient undergoing fibrinolysis has been well studied in many trials. In this study investigators will use clopidogrel or ticagrelor in randomized fashion to evaluate anti- platelet effect by measuring efficacy in vivo (pharmacodynamics) and blood levels of both drugs (Pharmacokinetics).

DETAILED DESCRIPTION:
This is an open label randomized pharmacodynamics study to compare platelet function reactivity of ticagrelor and clopidogrel after PCI in sub-set of patients who have undergone fibrinolysis at least 24 hour prior to PCI..A total of 70 patients will be enrolled. Prior to enrollment, patients have already undergone fibrinolysis (selected by the treating physician), aspirin (recommended dose 324 mg) on the first day and 81 mg daily thereafter, and Lovenox or heparin as per protocol of referring ER. Patients will undergo coronary angiography as standard of care and coronary stenting if indicated. Prior to angiography patient will be enrolled in this open label randomized protocol to receive clopidogrel or ticagrelor. Patients will be randomly assigned in a 1:1 ratio by open label study to receive either clopidogrel (Plavix, Sanofi-Aventis and Bristol-Myers Squibb; a 300-mg loading dose followed by 75 mg once daily) or ticagrelor (Brilinta, AstraZeneca; 180 mg loading and 90 mg twice daily) by a computerized system of randomization. Patients will receive clopidogrel or ticagrelor daily from enrollment to discharge. For patients who did not undergo PCI after enrollment, study drugs will be administered up to and including day 8th or hospital discharge, whichever comes first. Patients will be treated as per standard of care, and pharmacodynamics and pharmacokinetic study will be carried as per protocol. VerifyNow and VASP assay will be used to measure platelet reactivity for pharmacodynamic evaluation of ticagrelor vs Clopidogrel at specific time points: baseline (time 0), 30 mins, 1 hour, 2 hours, 8 hours and at 24 hours from first oral anti-platelet dose.. Blood will be collected from the sheath or ante-cubital vein into Vacutainer tubes for platelet function assay as below by VerifyNow and VASP. VerifyNow P2Y12 Assay: VerifyNow is a turbidimetric based system that measures platelet aggregation in the whole blood.8 This instrument measures an optical signal reported as P2Y12 Reaction Units (PRU). Vasodilator-Stimulated Phosphoprotein Phosphrylation (VASP) Assay: The measure of Vasodilator-Stimulated Phosphoprotein Phosphrylation (Biocytex Inc. Marseille, France), a method to quantify P2Y12 receptor reactivity, which reflects the extent of blockade of P2Y12 receptor blockade.9 Platelet reactivity index (PRI) is calculated by measuring VASP-P levels by mean fluorescence intensity (MFI) by stimulation with prostaglandin; PGE1and PGE1 plus ADP. PRI(%)=[(MFIPGE1)-(MFIPGE1+ADP)/(MFIPGE1)]×100%. ) Pharmacokinetic will be done at 30 min, 60 min, 120 min, 4 hours, 8 hours and at 24 hours. AUC from time 0-2 hours, Cmax at 2 hours, and Tmax at 2 hours for key secondary endpoint. Will collect Cmax and Tmax at all time points to be consistent, i.e. at 0, 30 min, 1 hour, 2 hour, 8 hours, and 24 hours when you draw PD measures at those time points and sample will be shipped.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 to 75 years of age
2. Ischemic discomfort lasting more than 20 mins at rest within 12 hours before randomization
3. ST-segment elevation of at least 0.1 mV in at least two contiguous limb leads, ST-segment elevation of at least 0.2 mV in at least two contiguous precordial leads, or left bundle-branch block that was not known to be old
4. Received fibrinolytic agent, an anticoagulant (if a fibrin-specific lytic agent was prescribed) and aspirin within 24-48 hours

Exclusion Criteria:

1. Hypersensitivity to ticagrelor or clopidogrel
2. Active Pathological Bleeding or history of intracranial bleeding
3. Concomitant use of oral anticoagulant
4. Concomitant use of 40 mg of Simvastatin or lovastatin
5. Concomitant strong CYP3A inhibitors such as ketoconazole, clarithromycin, nefazadone, ritonavir, atazanavir
6. Concomitant use of CYP2C19 inhibitors such as omeprazole or esomeprazole
7. Patients planned to urgent CABG
8. Thrombocytopenia
9. Dialysis
10. Use of oral antiplatelet agent (ticagrelor, prasugrel, Clopidogrel) within 7 days prior to enrollment
11. Use of GP IIb/IIIa inhibitors
12. Rescue PCI (PCI < 24 hours from symptom onset) -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01-02 (Estimated); Primary Completion 2015-05 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics (PRU and IPA) of ticagrelor vs Clopidogrel using VASP and VerifyNow | Change from baseline at 2 hours
  Pharmacodynamics at baseline, 30 min, 60 min, 120 min, 4 hours, 8 hours and at 24 hours

SECONDARY OUTCOMES:
Pharmacokinetic (AUC, Cmax, Tmax) | Change from baseline at 2 hours
  Pharmacokinetics at baseline, 30 min, 60 min, 120 min, 4 hours, 8 hours and at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh K Sharma, MD, FACC, FSCAI, FSCCT, Principal Investigator — Medical Center of South Arkansas
Locations (1):
- Medical Center of South Arkansas, El Dorado, Arkansas, United States